CLINICAL TRIAL: NCT07076667
Title: Comparative Effects of Benson's Relaxation Technique and Tai Chi in COPD
Brief Title: Effects of Benson's Relaxation and Tai Chi in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0353
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: Benson relaxation technique; Tai Chi; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benson'srelaxationtechnique (Active Comparator): "Benson's Relaxation Technique"along with the standard COPD care and medication.
  Interventions: Other: Benson's relaxation technique
- TaiChi (Experimental): "Tai Chi relaxation Technique" along with the standard COPD care and medication
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Benson's relaxation technique — effects of Benson's relaxation technique 5 days per week for 45 minutes for 8 weeks
  Arms: Benson'srelaxationtechnique
Other: Tai Chi — Tai Chi 5 days per week for 45 minutes for 8 weeks
  Arms: TaiChi

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive lung disorder that significantly impacts respiratory function and quality of life. As COPD patients often experience symptoms such as dyspnea, fatigue, and anxiety, non-pharmacological interventions like Benson's Relaxation Technique and Tai Chi are gaining attention for their potential benefits in managing these symptoms.This study aimed to compare the effectiveness of Benson's Relaxation Technique and Tai Chi on improving dyspnea, physical endurance, and quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common lung disease causing restricted airflow and breathing problems. An increasing number of studies show promising results for the performance of Tai Chi as an apppropriate addition in pulmonary rehabilitation. The Benson Relaxation Technique is a form of relaxation response therapy that can be beneficial for individuals with chronic obstructive pulmonary disease (COPD).This technique involves a series of steps designed to elicit the body's natural relaxation response, which can help manage stress and improve overall well-being. For COPD patients, incorporating breathing exercises can be especially beneficial. Slow,deep breathing can help improve oxygen intake and reduce the feeling of breathlessness. Controlled Breathing focus on taking slow, deep breaths in through the nose and out through the mouth. Pursed-lip breathing (breathing out through tightly pressed lips) can be particularly useful. It will be randomized clinical trial. Age of selected subjects will be between 40 to 60 years and data will be collected from Bahawalpur Victoria hospital. Sample size is 54. There will be 2 groups, group A will receive Benson'sr elaxation technique for 5 days per week for 45 minutes for 8 weeks and group B will receive TaiChi 5 days per week for 45 minutes for 8 weeks. Exercise will be performed to evaluate pulmonary functions and breathlessness. The Sampling Technique is non probability Convenience sampling technique. Study will be Conducted in Department of Pulmonary and Critical Care Medicine. After data collection, data will be analyzed by using SPSS version 25. It will be used aiming to determine the comparative effects of Benson's relaxation technique and Tai Chi in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age40 to 50
* Bothmaleandfemale
* DiagnosedmoderatetosevereCOPDpatients
* Participants must be physicallyable to participate in Tai Chi or Benson relaxation technique
* Participantsmustbewillingtoparticipate

Exclusion Criteria:

* Pulmonaryhypertension
* Congenitalheartdisease(recentmyocardialinfarction,unstableangina,or uncontrolled hypertension)
* Spinal deformities
* Lossof consciousness

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
MODIFIED BORG DYSPNEA SCALE | 8 weeks
  The MBS is a valid and reliable assessment tool for dyspnea. It is a tool to assess and rate the difficulty in breathing (dyspnea) rated from 0 to 10. 0 shows no dyspnea whereas 10 shows max dyspnea.
SIX MINUTE WALK TEST | 8 weeks
  The 6 MWT is safe,easy to administer,better tolerated, and reflects activities of daily living.When conducting the 6MWT do not walk with the patient and do not assist the patient in carrying or pulling his or her supplemental oxygen.The patient should walk alone,not with other patients.Do not use an oval or circular track. Use standardized phrases while speaking to the patient, because your encouragement and enthusiasm can make a difference of upto 30% in the 6MWD.Count the laps with a lap counter.
SPIROMETER | 8 weeks
  Spirometers arei nstruments to conduct spirometry tests.Earlier,spirometers were of either rolling model or bellows type but the recent ones are electronic and fully automated using digital turbine and flow sensors that require no calibration. Though spirometry does not measure the individual lung volumes,it measures the forced vital capacity (FVC).

SECONDARY OUTCOMES:
St.GEORGE'S RESPIRATORY QUESTIONNAIRE | 8 weeks
  The St George's Respiratory Questionnaire is a standardized self-completed questionnaire for measuring impaired health and perceived well-being ('quality of life') in airways disease. It has been designed to allow comparative measurements of health between patient populations and quantify changes in health following therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Iram Nawaz, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Bahawalpur Victoria Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavailles A, Brinchault-Rabin G, Dixmier A, Goupil F, Gut-Gobert C, Marchand-Adam S, Meurice JC, Morel H, Person-Tacnet C, Leroyer C, Diot P. Comorbidities of COPD. Eur Respir Rev. 2013 Dec;22(130):454-75. doi: 10.1183/09059180.00008612. PMID 24293462
- [Background] 2. LeungJM,ObeidatMe,SadatsafaviM,SinDD.Introductiontoprecisionmedicinein COPD. European Respiratory Journal. 2019;53(4).
- [Background] 3. AgustíA,VogelmeierC,FanerR.COPD2020:changesandchallenges.American Physiological Society Bethesda, MD; 2020. p. L879-L83.
- [Background] Nazari AM, Zare-Kaseb A, Arbabi Z, Gholampour MH, Emami Zeydi A, Ghazanfari MJ. The effect of Benson relaxation technique on cancer patients: a systematic review. Support Care Cancer. 2023 Nov 8;31(12):681. doi: 10.1007/s00520-023-08142-2. PMID 37938356
- [Background] JonesP,QuirkF,BaveystockC.TheStGeorge'sRespiratoryQuestionnaire.Respiratory medicine. 1991;85:25-31; discussion 3